CLINICAL TRIAL: NCT03630328
Title: Study of Angelica Gigas Dietary Supplements (Cogni.Q) and Potential Effects on Human Immune Cells
Brief Title: Angelica Gigas Dietary Supplements and Human Immune Cells
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Junxuan Lu, Professor of Pharmacology, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: STUDY00008009
Record Dates: First submitted 2018-08-09; First posted 2018-08-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Innate Immune Cells
Keywords: Cogni.Q; immune enhancement; natural killer cells; NK cells; Korean Angelica gigas; AGN

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cogni.Q (Experimental): 800 mg per day (Two 200 mg capsules in the morning and two 200 mg capsules in the evening) for 21 days
  Interventions: Dietary Supplement: Cogni.Q; Other: Placebo
- Placebo (Placebo Comparator): Two capsules in the morning and two capsules in the evening for 21 days
  Interventions: Dietary Supplement: Cogni.Q; Other: Placebo

INTERVENTIONS:
Dietary Supplement: Cogni.Q — AGN
Other: Placebo — Placebo

SUMMARY:
This human study will test the impact of dietary supplement vegicaps containing Korean Angelica root extract on 2 types of human immune cells: neutrophils that kill bacteria and other germs and natural killer (NK) cells that kill virus-infected cells and cancers. The investigators had done an earlier study with Korean Angelica supplement and discovered even a single dose of it increased blood neutrophils and NK cells within 24 h. In the new study, Korean Angelica capsules (Cogni.Q) will be compared head-to-head with dummy (placebo) capsules. This is to make sure the immune boosting actions are really from the Korean Angelica supplement.

ELIGIBILITY:
Inclusion Criteria:

* Subjects weighing between 110 to 240 pounds; their body mass index (BMI) should be in the range of 19 to 30
* Subjects having normal hepatic, renal function as assessed by history, physical and clinical chemistry analysis (CMP eGFR, see supporting document for normal reference ranges).
* Subjects with normal blood pressure (systolic below 120 mm Hg and diastolic below 80 mm Hg)

Exclusion Criteria:

* Subjects positive for HIV, HBV and HCV (self-reported)
* Subjects taking any kind of prescription medications regularly or within 10 days of the study will be excluded. Therefore, subjects with diabetes, major cardiovascular diseases, cancer, severe hypertension, severe hepatic cirrhosis or cirrhosis of the liver, and kidney disease (self-reported) will be excluded.
* Subjects using tobacco products, nicotine patches and excessive alcohol
* Subjects taking dietary or herbal supplements that contain AGN (e.g. Cogni.Q, Decursinol-50, Ache Action, Fast-Acting Joint Formula, EstroG-100/Profemin) within 10 days of the study.
* Non-English-speaking subjects

Ages: 21 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 40 (Estimated)
Dates: Start 2019-02-06 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Neutrophil counts and NK cell counts in peripheral blood | 70 days
  Using CBC diff to measure neutrophil counts, NK cells number will be enumerated using flowcytometer

SECONDARY OUTCOMES:
T cells in peripheral blood, | 70 days
  T cells number will be enumerated using flowcytometer
Plasma concentrations of pyranocoumarins, androgens, and inflammatory/anti-inflammatory cytokines. | 70 days
  Determine Plasma concentrations of pyranocoumarins (as compliance marker), androgens, and inflammatory/anti-inflammatory cytokines.
Lipid profiling | 70 days
  blood test will be done at every visit
NK mRNA signature | 70 days
  NK mRNA signature by RNA-seq transcriptomics using RNA prepared from Pax Gene tube-preserved whole blood collected on each visit
PBMC isolation for testing NK activity | 70 days
  PBMCs will be isolated at every blood draw and kept frozen. They will be used to determine NK cell activity in future.
CMP-EGFR | 70 days
  blood test will be done at every visit

CONTACTS AND LOCATIONS:
Overall Officials: Junxuan Lu, Ph.D., Principal Investigator — Penn State College of Medicine
Locations (1):
- Penn State College of Medicine, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-18): https://cdn.clinicaltrials.gov/large-docs/28/NCT03630328/Prot_SAP_000.pdf